CLINICAL TRIAL: NCT01496833
Title: Total Endovascular Aortic Arch Re-construction Study(TEARS)------China's Registry
Brief Title: Total Endovascular Aortic Arch Re-construction Study(TEARS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: XJ-20111126
Record Dates: First submitted 2011-12-13; First posted 2011-12-21 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Aorta Dissection; Aorta Aneurysm
Keywords: Aortic Diseases; Vascular Diseases; Cardiovascular Diseases; Treatment Outcome; Aorta Dissection; Aorta Aneurysm; Aorta pseudoaneurysm; Endovascular aortic repair
MeSH Terms: conditions — Aortic Dissection; Aortic Aneurysm; Aortic Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endovascular (Experimental): Total endovascular arch reconstruction
  Interventions: Device: Ankura Branched/Fenestrated Stent Graft

INTERVENTIONS:
Device: Ankura Branched/Fenestrated Stent Graft — Ankura Branched/Fenestrated Stent Graft（Lifetech Scientific Co.,LTD.，Shenzhen, China）
  Other Names: Ankura-TM Stent Graft; Ankura Branched Stent Graft; Ankura Fenestrated Stent Graft

SUMMARY:
The purpose of this study is to investigate the short to mid term efficacy and safety of a newly-developed branched stent graft in patients who had complex aortic lesions, such as ascending aortic/arch aneurysm, pseudo-aneurysm, Stanford Type A dissection, retrograde Stanford Type B dissection, dissection with primary tear located in the aortic arch, et al.

DETAILED DESCRIPTION:
Aneurysms and dissection involving the ascending aorta and aortic arch have historically been treated with open surgical techniques, requiring cardiopulmonary bypass and deep hypothermic circulatory arrest (DHCA). Despite increasing experience and refinement of these procedures, there remains a substantial rate of morality and morbidity. Total endovascular aortic arch and ascending aorta repair is one of the ultimate solutions of these diseases. However, this approach requires extensive technique and new device development. The goal of total endoluminal stent grafting is to re-construct the ascending aorta and aortic arch to cover the primary entry tear of the dissection and to remodel the aorta.Recently, branch and fenestrated stent-grafts has been developed to treat complex ascending and aortic arch disease, which was previously considered to be contraindicated for endovascular repair. This study aims to investigate the short to mid term efficacy and safety of a newly-developed branched stent graft in patients who had complex aortic lesions, such as ascending aortic/arch aneurysm, pseudo-aneurysm, Stanford Type A dissection, retrograde Stanford Type B dissection, dissection with primary tear located in the aortic arch, et al.

Primary outcome measure is all-cause mortality. Secondary outcome variables include conversion to stent and/or surgery, induced thrombosis of the false lumen, cardiovascular morbidity, aortic expansion (>5 mm/y of maximum diameter including true and false lumina), quality of life, and length of intensive care unit and hospital stay. The study designs to enroll 50 patients to be monitored for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Ascending aortic/arch aneurysm
2. Ascending aortic/arch pseudo-aneurysm
3. Stanford Type A dissection
4. Retrograde Stanford Type B dissection
5. Unclassified dissection with primary tear located in the aortic arch
6. Able to tolerate endotracheal intubation and general anesthesia
7. Subject's anatomy must meet the anatomical criteria to receive that implanted device
8. The subject or legal guardian understands the nature of the study and agrees to its provisions on a written informed consent form
9. Availability for the appropriate follow-up visits during the follow-up period
10. Capability to follow all study requirements

Exclusion Criteria:

1. ASA classification = V
2. Severe renal insufficiency defined as SVS risk renal status = 3
3. Severe respiratory insufficiency defined as SVS risk pulmonary status = 3
4. Presence of connective tissue disease
5. Active infection or active vasculitides
6. Pregnant woman or positive pregnancy test
7. Myocardial infarction or cerebrovascular accident within 6 weeks prior to study enrollment
8. Subject has had a cerebral vascular accident (CVA) within 2 months.
9. History of drug abuse
10. Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
11. Subject has a known allergy or intolerance to the device components.
12. Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.
13. Subject has a co-morbidity causing expected survival to be less than 1 year.
14. Enrolment in another clinical study
15. Unwillingness to cooperate with study procedures or follow-up visits

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
cumulative MACE (including death, rupture, paraplegia, aneurysm formation) | 12 months

SECONDARY OUTCOMES:
Endoleak | 12 months
  Endoleak of all types
Stent-graft migration/kinking | 12 months
  Stent-graft migration, stenosis, kinking and other conditions requiring re-intervention
cumulative cerebrovascular events | 12 months
  cumulative cerebrovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yang, MD,PhD, Principal Investigator — Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University; Dinghua Yi, M.D., PhD., Study Chair — Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University
Locations (1):
- Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China